CLINICAL TRIAL: NCT06123286
Title: An Open Label, Randomized, Waitlist Controlled Trial of Tart Cherry and Omega-3's for Aromatase Inhibitor Musculoskeletal Symptoms
Brief Title: Tart Cherry and Omega-3's for Aromatase Inhibitor Musculoskeletal Symptoms
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Philip Chang (Other)
Collaborators: The Cherry Marketing Institute (Unknown)
Responsible Party: Sponsor-Investigator, Philip Chang, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2022-08-CHANG-TaCO3AIMSS
Record Dates: First submitted 2023-10-16; First posted 2023-11-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Aromatase Inhibitor Associated Musculoskeletal Symptoms (AIMSS); Joint Pain
Keywords: Aromatase Inhibitor Therapy; AIMSS; Aromatase Inhibitor Associated Musculoskeletal Symptoms (AIMSS); Tart Cherry; Omega 3 Fatty Acids Fish Oil; Female Breast Cancer; Aromatase Inhibitor Arthralgia
MeSH Terms: conditions — Breast Neoplasms; Arthralgia | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 : Wait list control (No Intervention): No supplement but will be offered supplements after finishing the study
- Group 2 : Tart Cherry and Omega 3 FA (Fish Oil) (Experimental)
  Interventions: Drug: Tart Cherry; Drug: Omega 3 FA (Fish Oil)

INTERVENTIONS:
Drug: Tart Cherry — 1 ounce of Tart Cherry Concentrate (King Orchard) mixed with 8 ounces of water daily for 12 weeks
  Arms: Group 2 : Tart Cherry and Omega 3 FA (Fish Oil)
Drug: Omega 3 FA (Fish Oil) — 2 capsules of Omega 3 FA (Fish Oil) (Nordic Naturals Ultimate Omega) [650 mg EPA and 450 mg DHA per capsule] daily for 12 weeks
  Arms: Group 2 : Tart Cherry and Omega 3 FA (Fish Oil)

SUMMARY:
Both Tart Cherry and Omega 3 FAs have better side effect profiles compared to other commonly used medications for AIMSS, such as nonsteroidal anti-inflammatories, steroids, and serotonin norepinephrine reuptake inhibitors. Additionally, in our clinics we often find that patients tend to be more receptive to taking a supplement as opposed to an additional medication. Further, both Tart Cherry concentrate and fish oil have beneficial properties for helping with joint stiffness in general, in addition to other health issues like insomnia.

There is preliminary evidence in mouse models that when given together, these supplements may have an even greater anti-inflammatory effect than when taken separately14. Although to our knowledge, no human studies have tested this hypothesis. This study has been designed to test the hypothesis that Tart Cherry and fish oil when given in combination over a 12-week period could produce beneficial changes in joint function when compared to Tart Cherry or fish oil in isolation in an obese breast cancer population experiencing AIMSS. Secondary outcomes to be assessed include pain, functional performance, quality of life and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis (Stage I-III) with any hormonal status.
* Females aged ≥ 18 years.
* Currently receiving AI therapy.
* BMI ≥ 27.
* Clinical diagnosis of AIMSS.
* Omega-3 Index <8%.
* Average joint pain score ≥ 4 on the Brief Pain Inventory (BPI) within 7 days of enrollment.
* Written informed consent obtained from subject and ability and willingness of subject to comply with the requirements of the study.

Exclusion Criteria:

* Current use of anticoagulant medications (Including but not limited to Warfarin, Lovenox, Eliquis, Xarelto).
* Allergy to cherries or fish/fish products.
* Lifetime history of rheumatoid arthritis and/or inflammatory joint diseases (Including but not limited to reactive arthritis, ankylosing spondylitis, and psoriatic arthritis).
* Uncontrolled diabetes mellitus as determined by treating physician (with or without the use of glucose lowering medications and/or insulin).
* Lifetime history of stroke or transient ischemic attacks.
* New use or dose change of oral or topical analgesics in the previous 14 days. (Including but not limited to opioids, non-steroidal anti-inflammatories, acetaminophen, SNRI's, SSRI's, gabapentinoids, tricyclic antidepressants, and muscle relaxants).
* Oral or intra-articular steroid use in the previous 30 days (Including but not limited to dexamethasone, prednisone, methylprednisolone, triamcinolone, hydrocortisone).
* History of joint fracture or surgery of the symptomatic joint in the previous 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess changes in joint function between groups. | 6 Months
  Changes in joint symptoms will be assessed via the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC Pain score ranges from 0% to 100% with higher scores indicating greater difficulty with activities of daily living.

SECONDARY OUTCOMES:
To assess changes in nociplastic pain between groups. | 6 Months
  Changes in nociplastic pain will be measured by composite score on Symptom Severity Scale. The Symptom Severity Scale ranges from 0-12 with higher scores equating to increased nociplastic pain.
To assess changes in nociplastic pain between groups. | 6 Months
  Changes in nociplastic pain will be measured by composite score on Widespread Pain Index. The Widespread Pain Index score ranges from 0-19 with higher scores equating to increased nociplastic pain.
To assess changes in functional performance between groups. | 6 Months
  Functional Performance will be measured by changes in the Patient-Reported Outcomes Measurement Information System (PROMIS) Cancer 3D Function Profile. The PROMIS Cancer 3D Function Profile has 3 subgroups including Physical Function, Fatigue and Social Participation. The Physical Function score ranges from 5-30 with higher scores equating to better function. The Fatigue score ranges from 3-15 with higher scores equating to less fatigue. The Social Participation score ranges from 3-15 with higher scores equating to worse social participation.
To assess changes in quality of life between groups. | 6 Months
  Quality of Life will be measured by changes in the Patient-Reported Outcomes Measurement Information System (PROMIS) PROMIS-29+2. The PROMIS-29+2 has 8 subgroups including physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles, pain interference and cognitive function. All subgroups are scored from 4-20 except for cognitive function which is scored from 2-10.
To assess changes in cognition between groups. | 6 Months
  Cognition will be measured by changes in the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function 8a Short Form. The PROMIS Cognitive Function Short Form 8a score ranges from 8 to 40 with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chang, DO, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - CS Cancer at the Hunt Cancer Center, Torrance, California

IPD SHARING:
Plan to Share IPD: No